CLINICAL TRIAL: NCT02022683
Title: A Multi-center, Prospective, Randomized, Controlled Trial of Endobronchial Valve Therapy vs. Standard of Care in Heterogeneous Emphysema
Brief Title: To Improve Lung Function and Symptoms for Emphysema Patients Using Zephyr Valves
Acronym: TRANSFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 630-0015/A
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: COPD; Heterogeneous Emphysema
Keywords: Endoscopic lung volume reduction; Endobronchial valves
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic Lung Volume Reduction (Experimental): Patients are implanted with Zephyr Valves
  Interventions: Device: ELVR (Endoscopic Lung Volume Reduction) with Zephyr Valves
- Standard of Care (No Intervention): Patients are given Standard Medical Care

INTERVENTIONS:
Device: ELVR (Endoscopic Lung Volume Reduction) with Zephyr Valves
  Arms: Endoscopic Lung Volume Reduction

SUMMARY:
To compare the clinical outcomes of Endoscopic Lung Volume Reduction (ELVR) using Pulmonx Zephyr Valves vs. Standard of Care (SoC) in the treatment of heterogeneous emphysema subjects in a controlled trial design setting.

ELIGIBILITY:
Inclusion Criteria:

1. Obtained informed consent.
2. Diagnosis of heterogeneous emphysema with a heterogeneity index of ≥10 % between target and adjacent lobes.
3. Subjects of both genders of at least 40 years of age.
4. 15 % predicted ≤ FEV1≤ 45% predicted.
5. TLC > 100% and RV ≥ 180% predicted.
6. 150 meters < 6MWD < 450 meters.
7. Non-smoker >8 weeks prior to signing the Informed Consent.
8. CV negative target lobe.

Additional inclusion criterion French CIP*:

- If treated in France, Subject must be entitled to French social security

Exclusion Criteria:

1. Any contraindication for bronchoscopic procedure.
2. Evidence of active pulmonary infection.
3. History of 2 or more exacerbations requiring hospitalization over the past 12 months.
4. Known pulmonary hypertension that according to the physician will be unsuitable for EBV treatment.
5. Myocardial infarction or other relevant cardiovascular events in the past 6 months.
6. Significant bronchiectasis seen at CT scan.
7. Greater than two tablespoons of sputum production per day.
8. Prior LVR or LVRS procedure. Criterion 8 French CIP wording*: Prior lung transplant, median sternotomy, LVR or LVRS procedure (including lobectomy).
9. Pulmonary nodule requiring follow-up within any lobe.
10. Pregnant or nursing women. French CIP wording*: Subject is pregnant or lactating, or plans to become pregnant within the study timeframe.
11. Hypercapnia (paCO2 > 7.33 kPa).
12. Current diagnosis of asthma.
13. > 25mg Prednisolon (or equivalent) use/days.
14. Any other condition that as judged by the investigator may make follow-up or investigations inappropriate.
15. Evidence of pleural adhesions or earlier pulmonary surgery.
16. Severe Bullous Emphysema (> 1/3 Hemithorax)
17. Any subject that according to the Declaration of Helsinki is unsuitable for enrollment.

Additional exclusion criteria in the French CIP*:

* History of allergy to silicone and/or nitinol.
* If treated in France, Subject is a "personne vulnerable" as defined by French regulation.
* Simultaneous participation in another drug and/or medical device related clinical.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1-second (FEV1) - Responders | Between baseline and 3 months
  The percentage of trial participants in the EBV treatment arm meeting the minimally clinically important difference (MCID) of >12% improved forced expiratory volume in one second (FEV1), obtained immediately following bronchodilator therapy, as compared to the percentage in the control arm at 3 months post-procedure.

SECONDARY OUTCOMES:
St George's Respiratory Questionnaire (SGRQ) - Absolute change | Between Baseline and 3, 6, 12, 18 and 24 months
  Absolute change in the SGRQ in the EBV treatment arm at 3, 6, 12, 18 and 24 months relative to Baseline and the difference between the two arms at 3, 6 and 12 months.
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts:
  Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease)
  A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations.
St George's Respiratory Questionnaire (SGRQ) - Percent change | Between Baseline and 3, 6, 12, 18 and 24 months
  Percent change in the SGRQ in the EBV treatment arm at 3, 6, 12, 18 and 24 months relative to Baseline and the difference between the two arms at 3, 6 and 12 months.
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts:
  Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease)
  A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations.
St George's Respiratory Questionnaire (SGRQ) - Responders | Between Baseline and 3, 6, 12, 18 and 24 months
  Percentage of subject achieving the MCID for SGRQ in the EBV treatment arm at 3, 6, 12, 18 and 24 months, compared to SoC at 3, 6 and 12 months.
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts:
  Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease)
  A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations.
6-minute walk distance (6MWT) - Absolute change | Between Baseline and 3, 6, 12, 18, 24 months
  Absolute change in 6MWD in the EBV treatment arm at 3, 6, 12, 18, 24 months relative to Baseline and the difference between the two arms at 3, 6 and 12 months.
6-minute walk distance (6MWT) - Percent change | Between Baseline and 3, 6, 12, 18, 24 months
  Percent change in 6MWD in the EBV treatment arm at 3, 6, 12, 18, 24 months relative to Baseline and the difference between the two arms at 3, 6 and 12 months.
6-minute walk distance (6MWT) - Responders | Between Baseline and 3, 6, 12, 18, 24 months
  Percentage of subject achieving the MCID for 6MWD in the EBV treatment arm at 3, 6, 12, 18 and 24 months, compared to SoC at 3, 6 and 12 months.
Forced Expiratory Volume in 1-second (FEV1) - Absolute change | Between Baseline and 3, 6, 12, 18, 24 months
  Absolute change in FEV1 in the EBV treatment arm at 3, 6, 12, 18, 24 months relative to Baseline and the difference between the two arms at 3, 6 and 12 months.
Forced Expiratory Volume in 1-second (FEV1) - Percent change | Between Baseline and 6, 12, 18 and 24 months
  Percentage of subject achieving the MCID for FEV1 in the EBV treatment arm at 6, 12, 18 and 24 months, compared to SoC at 6 and 12 months.
Forced Expiratory Volume in 1-second (FEV1) - Responders | Between Baseline and 3, 6, 12, 18, 24 months
  Absolute change in FEV1 in the EBV treatment arm at 3, 6, 12, 18, 24 months relative to Baseline and the difference between the two arms at 3, 6 and 12 months.
mMRC (Modified Medical Research Council) score - Responders | Between Baseline and 3, 6, 12, 18 and 24 months
  Percentage of subject in the EBV treatment arm achieving the MCID for the Modified Scale Research Council Dyspnea Score (mMRC) at 3, 6, 12, 18 and 24 months and the difference between the two arms at 3, 6 and 12 months.
  The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations.
Target Lobar Volume Reduction (TLVR) - Absolute change | Between baseline and 45 days
  Absolute change in target lobe volume at 45 days in the EBV treatment arm relative to Baseline as assessed by quantitative HRCT analysis (TLVR: Target Lobar Volume Reduction).
Target Lobar Volume Reduction (TLVR) - Percent change | Between baseline and 45 days
  Percent change in target lobe volume at 45 days in the EBV treatment arm relative to Baseline as assessed by quantitative HRCT analysis (TLVR: Target Lobar Volume Reduction).
Target Lobar Volume Reduction (TLVR) - Responders | Between baseline and 45 days
  Percentage of subjects in EBV arm with a TLVR > 350ml at 45 days relative to baseline.

OTHER OUTCOMES:
Adverse Events | Between baseline and 24 months
  Adverse events (condition/procedure related AE's, SAE's, ADE's and SADE's) occurring up to 24 months post EBV placement and up to 12 months post randomization (for any remaining subjects in the SoC group).
PaO2 - Absolute change | Between baseline and 3 months
  Absolute change in PaO2 in the EBV treatment arm at 3 months relative to Baseline.
PaO2 - Percent change | Between baseline and 3 months
  Percent change in PaO2 in the EBV treatment arm at 3 months relative to Baseline.
Residual Volume (RV) - Absolute change | Between Baseline and 3, 6 and 12, 18 and 24 months
  Absolute change in residual volume (RV) in the EBV treatment arm at 3, 6 and 12, 18 and 24 months relative to Baseline and the difference between the two arms at 3, 6 and 12 months.
Residual Volume (RV) - Percent change | Between Baseline and 3, 6 and 12, 18 and 24 months
  Percent change in residual volume (RV) in the EBV treatment arm at 3, 6 and 12, 18 and 24 months relative to Baseline and the difference between the two arms at 3, 6 and 12 months.
EQ-5D Summary Index - Absolute change | Between Baseline and 3, 6, 12, 18 and 24 months
  Absolute change relative to Baseline in the EBV treatment arm at 3, 6, 12, 18 and 24 months of the EQ-5D Summary Index and the difference between the two arms at, 3, 6 and 12 months.
  EQ-5D is a standardized instrument used to measure health-related quality of life for a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
EQ-5D Summary Index Percent change | Between Baseline and 3, 6, 12, 18 and 24 months
  Percent change relative to Baseline in the EBV treatment arm at 3, 6, 12, 18 and 24 months of the EQ-5D Summary Index and the difference between the two arms at, 3, 6 and 12 months.
  EQ-5D is a standardized instrument used to measure health-related quality of life for a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
Mean number of additional hospitalizations and/or visits caused by respiratory conditions | Between baseline and 24 months
  The mean number of visits (Number of participants reporting visits/total number of visits) caused by respiratory conditions during the study period will be recorded for health economical purposes in both treatment and control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Hillerdal, MD, PhD, Principal Investigator — Uppsala University Hospital, Sweden
Locations (17):
- Belgium (2):
  - Universiteit Gent, Ghent
  - AZ Delta, Menen
- France (4):
  - CHU, Grenoble
  - CHU Hôpital Pasteur, Nice
  - Groupe Hospitalier Pitié Salpétrière, Paris
  - Hôpital Bichat Claude Bernard, Paris
- Germany (3):
  - Charité Campus Virchow-Klinikum, Berlin
  - Ruhrlandklinik Westdeutsches Lungenzentrum, Essen
  - Thoraxklinik am Universitäts Klinikum Heidelberg, Heidelberg
- University Medical Center Groningen, Groningen, Netherlands
- Sweden (2):
  - Skane University Hospital, Lund
  - Uppsala University Hospital, Uppsala
- United Kingdom (5):
  - Sherwood Forest Hospitals NHS, Sutton in Ashfield, Nottinghamshire
  - West of Scotland Regional Heart & Lung Centre - Golden Jubilee National Hospital, Clydebank, West Dunbartonshire Scotland
  - University Hospital of Wales, Cardiff
  - The Royal Brompton Hospital & Harefield NHS Foundation Trust, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bakker JT, Hartman JE, Klooster K, Charbonnier JP, Tsiaousis M, Vliegenthart R, Slebos DJ. Endobronchial valve treatment improves chest-CT diaphragm configuration in COPD. Respir Med. 2024 Nov-Dec;234:107856. doi: 10.1016/j.rmed.2024.107856. Epub 2024 Nov 6. PMID 39515624
- [Derived] Kemp SV, Slebos DJ, Kirk A, Kornaszewska M, Carron K, Ek L, Broman G, Hillerdal G, Mal H, Pison C, Briault A, Downer N, Darwiche K, Rao J, Hubner RH, Ruwwe-Glosenkamp C, Trosini-Desert V, Eberhardt R, Herth FJ, Derom E, Malfait T, Shah PL, Garner JL, Ten Hacken NH, Fallouh H, Leroy S, Marquette CH; TRANSFORM Study Team *. A Multicenter Randomized Controlled Trial of Zephyr Endobronchial Valve Treatment in Heterogeneous Emphysema (TRANSFORM). Am J Respir Crit Care Med. 2017 Dec 15;196(12):1535-1543. doi: 10.1164/rccm.201707-1327OC. PMID 28885054